CLINICAL TRIAL: NCT03324659
Title: Combined Meditation and Exercise as a Treatment for Patients With Chronic Back Pain
Brief Title: Meditation and Exercise to Treat Chronic Back Pain
Acronym: MedExT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Matthew Kostek, Assistant Professor, Duquesne University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol50
Record Dates: First submitted 2017-10-17; First posted 2017-10-30 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Chronic Low Back Pain
Keywords: Mindfulness; Exercise; Meditation; Back pain
MeSH Terms: conditions — Motor Activity; Back Pain | interventions — Exercise; Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Meditation (Experimental): The Exercise and Meditation group will practice mindfulness meditation immediately before walking treadmill exercise, five days per week for four weeks.
  Interventions: Behavioral: Exercise and Meditation
- Control (Sham Comparator): The Control group will listen to an audio book followed by quiet rest, five days per week for four weeks.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Exercise and Meditation — The Exercise and Meditation group will listen to recorded meditations (15 minutes) that are based on mindfulness. They will then walk on a treadmill for 30 minutes at a moderate intensity. The intervention is completed five days per week for four weeks.
  Arms: Exercise and Meditation
Behavioral: Control — The Control group will listen to a recorded audio book for 15 minutes, They will then sit quietly for 30 minutes. The intervention is completed five days per week for four weeks.
  Arms: Control

SUMMARY:
This study evaluates the analgesic effect of a combination treatment of exercise and mindfulness based meditation in patients with chronic back pain. Half of the participants will partake in a 4-week exercise and meditation intervention, while the other half will receive a placebo treatment. The investigators hypothesize that a combination treatment reduces disability and pain more than the control intervention.

DETAILED DESCRIPTION:
Exercise and mindfulness based mediation can both produce analgesic effects in patients with chronic pain, but the mechanisms are not clear.

Combining treatments could produce analgesic effects that are additive, synergistic, or counteractive to each other. Here, the investigators examine the effects of a 4-week intervention in patients with chronic low back pain. Patients are assigned to a meditation/exercise group or a control group. The investigators will measure pain and disability using a variety of tools including surveys (disability, anxiety, mindfulness, and pain), pain VAS scales, and quantitative sensory testing.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of clinically diagnosed nonspecific low back pain for at least 6 months
2. Body mass index within the normal to overweight range (18.5-29.9)
3. Resting heart rate 60 to 100 beats per minute
4. Resting blood pressure less than or equal to 140/90
5. Able to independently ambulate community distances without external support (e.g., walker, cane)

   Exclusion Criteria:
6. Age less than 18 or greater than 60 years
7. BMI ≥ 30 or ≤ 18.4
8. Cardiovascular or respiratory disease
9. Neurological disease, unrelated to low back pain
10. Radicular low back pain
11. Back pain associated with neuropathy
12. Diabetes mellitus, Types 1 and 2
13. Diagnosed with a chronic pain condition, unrelated to low back pain
14. Acute pain
15. Regular participation in high intensity athletic/sporting activities
16. Sedentary lifestyle
17. Currently pregnant
18. Current cigarette smoker
19. On-going litigation associated with back pain
20. Inability to walk independently without external support (e.g. walker).
21. Regular participation in meditation techniques or training in Mindfulness-based stress reduction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Roland Morris Disability Questionnaire | baseline and 4 weeks
  The Roland-Morris Disability Questionnaire is designed to assess self-rated physical disability caused by low back pain. The patient is asked to tick a statement when it applies to him that specific day, this makes it possible to follow changes in time. The end score is the sum of the ticked boxes. The score ranges from 0 (no disability) to 24 (max. disability).

SECONDARY OUTCOMES:
Change in Cutaneous Sensation | baseline and 4 weeks
  Subjects will be examined using cutaneous sensory filaments on the forearm with data recorded in grams.
Fear Avoidance Beliefs Questionnaire | baseline and 4 weeks
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a questionnaire based on the Fear-Avoidance Model of Exaggerated Pain Perception, a model created in attempts to explain why some patients with acute painful conditions can recover while other patients develop chronic pain from such conditions. The FABQ measures patients' fear of pain and consequent avoidance of physical activity because of their fear. This questionnaire consists of 16 items, with each item scored from 0-6. Higher scores on the FABQ are indicative of greater fear and avoidance beliefs
Freiburg Mindfulness Inventory | baseline and 4 weeks
  The FMI is a 14-item questionnaire for measuring mindfulness. It is most suitable in generalized contexts, where knowledge of the Buddhist background of mindfulness cannot be expected. The 14 items cover all aspects of mindfulness. The purpose is to characterize the experience of mindfulness. The subject is asked to answer every statement as honestly and spontaneously as possible. Each statement is scored on a 1 to 4 scale and a composite score is calculated from all statements.
VAS back pain (intensity & unpleasantness) | baseline, daily (pre and post intervention), and 4 weeks
  Participants will be asked to rate their current level of back pain intensity on a Visual Analog Scale (VAS) ranging from 0 to 10
State-Trait Anxiety Inventory (STAI) | baseline and 4 weeks
  The STAI is an introspective psychological inventory consisting of 40 self-report items pertaining to anxiety affect. It distinguishes between a person's state and trait anxiety levels. The A-Trait and A-State scales comprise 20 items each, scored on a 4-point Likert-type response scale. Higher STAI scores suggest higher levels of anxiety.
Change in Pressure Sensation | baseline and 4 weeks
  Subjects will be examined using a pressure algometer to determine a pressure pain threshold, measured in Newtons
Change in Heat unpleasantness | baseline and 4 weeks
  Subjects will be examined using a heat block with a determined temperature threshold. Subjects will report unpleasantness using a VAS scale.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C. Kostek, PhD, Principal Investigator — Duquesne University; Benedict J Kolber, PhD, Principal Investigator — Duquesne University; Eric Helm, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT03324659/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT03324659/SAP_002.pdf